CLINICAL TRIAL: NCT04237259
Title: Traditional Chinese Medicine (TCM) Pediatric Massage for the Treatment of Attention Deficit Hyperactivity Disorder (ADHD) Symptoms in Preschool Children: A Pilot Randomized Controlled Trial
Brief Title: Traditional Chinese Medicine Pediatric Massage for Attention Deficit Hyperactivity Disorder Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YEUNG Wing Fai, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCM ped msg_ADHD
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent-administered TCM massage group (Experimental): Parents of subjects in the parent-administered TCM massage group (n=30) will attend 2 training sessions (5 hours in total) to learn and practice the parent-administered TCM massage for ADHD before treatment starts. The parents will be told to practice the TCM massage on their child every 2 days for 2 months.
  Interventions: Other: Parent-administered TCM pediatric massage training
- Parent-child interaction group (Active Comparator): Parents in the parent-child interaction group (comparison group, n=30) will attend a 3-hour training course on line and spend extra time on interacting with their child at home.
  Interventions: Other: Progressive Muscle Relaxation Exercise

INTERVENTIONS:
Other: Parent-administered TCM pediatric massage training — Massage therapy is a kind of complementary and alternative therapy, which involves a number of techniques such as friction, pressing, rubbing, grasping, pinching, and kneading. TCM pediatric massage, also called pediatric tuina and pediatric anmo, is a special part of TCM massage system that usually use lines or surfaces rather than points as acupoints and the manipulations are different from those of TCM adult massage. From TCM perspective, the pathogenesis of ADHD is the abnormal exuberance of yang, which can be relieved by specific approaches of massage.
  Participants in this group will receive two TCM pediatric massage training sessions (5 hours in total, one is 3 hours, and the other is 2 hours). The protocol will be tested for feasibility at the first feasibility stage (the first 8 subjects).
  Arms: Parent-administered TCM massage group
Other: Progressive Muscle Relaxation Exercise — The principle of progressive muscle relaxation exercise is to achieve a relaxation state through relaxing our muscles. With training, we become more familiarized with the sense of relaxation so that we can voluntarily induce this sensation in the face of a stressor.
  Arms: Parent-child interaction group

SUMMARY:
This project is designed to preliminarily assess the effects and feasibility of parent-delivered TCM pediatric massage for ADHD symptoms in preschool children.

DETAILED DESCRIPTION:
Objectives: To preliminarily assess the effects and feasibility of parent-delivered TCM pediatric massage for ADHD symptoms in preschool children.

Hypothesis: The parent-delivered TCM pediatric massage group would have greater improvement in children's hyperactivity, anxiety, and sleep disturbance symptoms when compared to the parent-child interaction group.

Design and subjects: In this pilot randomized controlled trial, 60 pair of children with pre-specified ADHD symptoms and their parent will be recruited and randomized to parent-administered TCM pediatric massage comparison group, and parent-child interaction group at a 1: 1 ratio.

Interventions: Parents of subjects in the parent-administered TCM massage group (n=30) will attend 2 training sessions (5 hours in total) to learn and practice the parent-administered TCM massage for ADHD before treatment starts. The parents will be told to practice the TCM massage on their child every 2 days for 2 months. Parents in the parent-child interaction group (comparison group, n=30) will attend a 3-hour training course on line and spend extra time on interacting with their child at home.

Main outcome measures: The primary outcome measure is the Swanson, Nolan and Pelham Parent Scale (SNAP-IV-P). Other outcomes include Preschool Anxiety Scale (PAS), Children's Sleep Habits Questionnaire (CSHQ), Parental Stress Scale (PSS) for parental stress, and the Clinical Global Impression (CGI).

Data Analysis: Differences in the scale scores and test parameters between groups will be examined using a linear mixed-effects model.

Expected results: Subjects in the parent-administered TCM massage group will have greater improvements in the ADHD symptoms compared to those in the parent-child interaction group at week 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the children are:

1. children between 3-7 years old by the time of the start of the assessment;
2. having a score equal to or higher than the borderline cutoff of the Strengths and Weaknesses of ADHD Symptoms and Normal Behaviors Rating Scale (SWAN), indicating the children had moderate ADHD symptoms.

The children with ADHD symptoms of hyperactivity, anxiety, or inattention will be recruited in this study. The rationale for not restricting the study to children with formal diagnosis is that many children are first assessed by professionals after 7 years old, and therefore many children with severe hyperactivity, anxiety, and sleep disturbance symptoms have not yet received a diagnosis. For these children, they together with their parents should be considered according to the inclusion criteria.

Inclusion criteria for parents are:

1. able to communicate using Mandarin;
2. willing to learn the knowledge and manipulations of TCM pediatric massage for treating ADHD;
3. available to take their child to hospital for treatment and conduct manipulations at home according to the study process;
4. agree to give informed consent.

Exclusion Criteria:

Exclusion criteria for children are:

1. currently receiving other massage therapy;
2. having other developmental disability such as autism spectrum disorders or intellectual disability;
3. having acute infection diseases (such as scarlet fever, chickenpox), hemorrhagic diseases (like bleeding, local places of various kinds of malignant tumor), or dermatological problems (e.g. scald, severe skin lesion, or skin infections);
4. having any severe illness or medical condition that the investigator deems not appropriate to receive TCM massage (e.g. bone fractures and paraplegia).

Exclusion criteria for parents are:

1. having any severe psychiatric disorder, such as major depressive disorder;
2. having difficulties to conduct massage therapy due to physical problems;
3. having a score of Montreal Cognitive Assessment (MoCA) less than 22, indicating cognitive impairment (Appendix 1: Montreal Cognitive Assessment (MoCA) - Chinese Version)

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in The self-completed Swanson, Nolan and Pelham Parent Scale (SNAP-IV-P) - ADHD Scale | Baseline, week 4, week 8
  It has 26 items that include 18 ADHD symptoms (nine inattentive, nine hyperactive or impulsive) and as specified in the DSM-5. Items are rated for frequency by the parent or teacher on a 4-point scale (0 = not at all to 3 = very much) and average ratings per item are then calculated for each subscale.

SECONDARY OUTCOMES:
Preschool Anxiety Scale (PAS) | Baseline, week 4, week 8
  The PAS-SC is a 34-item parent-rated scale, which assesses anxiety symptoms in young children across six subscales: panic attack and agoraphobia, separation anxiety, physical injury fears, social phobia, obsessive compulsive, generalized anxiety disorder/overanxious disorder.
Children's Sleep Habits Questionnaire (CSHQ) | Baseline, week 4, week 8
  CSHQ is a retrospective, 33- item parent questionnaire that has been used in a number of studies to examine sleep behaviour in young children.
Parental Stress Scale (PSS) | Baseline, week 4, week 8
  PSS is a measure of "individual differences in the level of stress associated with raising children'', which consists of 18 items on the perception of parental stress and uses a Likert style rating scale.
Clinical Global Impression (CGI) | Baseline, week 4, week 8
  The CGI is usually used as a standard primary measure in studies investigating the efficacy of pharmacological treatments for psychiatric conditions such as depression, social anxiety disorder, panic disorder and bipolar disorder.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen SC, Yu J, Suen LK, Sun Y, Pang YZ, Wang DD, Zhao WX, Yeung WF. Pediatric tuina for the treatment of attention deficit hyperactivity disorder (ADHD) symptoms in preschool children: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2020 Nov 5;6(1):169. doi: 10.1186/s40814-020-00704-z. PMID 33292826